CLINICAL TRIAL: NCT05975372
Title: Blossom® Smart Expander Device for Tissue Expander/Implant-Based Breast Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Marz Medical, Inc. (Unknown)
Responsible Party: Principal Investigator, Dung Nguyen, Clinical Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 67363
Record Dates: First submitted 2023-07-27; First posted 2023-08-03 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-07

CONDITIONS: Tissue Expansion; Implant Based Breast Reconstruction
Keywords: Implant based breast reconstruction; Tissue expansion

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either undergo tissue expansion with the Blossom device (intervention group) or standard tissue expansion methods (control group).
Who Masked: Outcomes Assessor
Masking Description: By nature of the visible device, participants and care providers cannot be blinded to the treatments. Analysis of data generated during the trial will be blinded to the treatment groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Blossom tissue expander (Experimental): The intervention group involves the placement of the Mentor Spectrum tissue expander coupled with Blossom Syringe Assist device inserted above the pectoralis major muscle in the usual fashion. The nature of the surgery remains identical to that employed for conventional breast tissue expander insertion for reconstruction or augmentation.
  Postoperative follow-up will occur within 1 week of surgery. Weekly follow-ups with documentation of clinical data throughout will also take place until completion of the expansion, stabilization of surgical scars, and removal of all percutaneous drains. Tissue expansion will be automatic via the Blossom device until appropriate volume is achieved. Thereafter, follow-ups will be scheduled as needed (monthly) according to usual clinical practice in implant-based breast reconstruction in preparation for the second stage expander to definitive implant exchange.
  Interventions: Device: Blossom tissue expander
- Standard tissue expansion (Active Comparator): The standard tissue expansion group will undergo the same procedure with placement of the Mentor Spectrum tissue expander inserted above the pectoralis major muscle in the usual fashion. Postoperative follow-up will occur within 1 week of surgery. Weekly follow-ups with documentation of clinical data throughout will also take place until completion of the expansion, stabilization of surgical scars, and removal of all percutaneous drains. Tissue expansion will be achieved via serial injections of sterile saline into the tissue expander during postoperative follow up visits. Thereafter, follow-ups will be scheduled as needed (monthly) according to usual clinical practice in implant-based breast reconstruction in preparation for the second stage expander to definitive implant exchange. The postoperative follow-up and subsequent surgery to exchange the device to a permanent implant is normal part of standard care.
  Interventions: Device: Standard tissue expansion

INTERVENTIONS:
Device: Blossom tissue expander — Mentor spectrum adjustable saline breast implant for expansion is placed with the Blossom tissue expander above pectoralis major during first stage surgery of an implant-based breast reconstruction/ augmentation.
  Other Names: Blossom smart expander device; Marz blossom syringe assist device; Blossom syringe assist device
  Arms: Blossom tissue expander
Device: Standard tissue expansion — Mentor spectrum adjustable saline breast implant for expansion is placed with (without the Blossom tissue expander) above pectoralis major during first stage surgery of an implant-based breast reconstruction/ augmentation.
  Arms: Standard tissue expansion

SUMMARY:
The conventional breast tissue expander used for breast reconstruction/ augmentation requires weekly or biweekly injections of saline through the skin and into an integrated port in the implant using a needle and syringe in order to expand breast skin, which is an in-office procedure and can be uncomfortable for patients. Blossom Smart Expander Technology, currently available on the market, aims to achieve the same tissue expansion while avoiding frequent injections through the skin by means of an expansion device that slowly and continuously injects a very small amount of saline. Expansion of the device is based on pressure and volume in the expander, allowing for a tailored expansion process for individual patients' physiology. The purpose of this study is to assess the clinical effectiveness of Blossom Smart Expander Technology in 2-staged tissue expander/implant-based breast reconstruction/ augmentation compared to standard tissue expansion methods.

DETAILED DESCRIPTION:
All consenting patients presenting to Dr. Dung Nguyen's breast reconstruction clinic and opting for 2-staged tissue expander/implant-based breast reconstruction or augmentation will be given the option of study enrollment. Consenting patients will be enrolled and randomized 1:1 to undergo standard 2-staged breast reconstruction/ augmentation with conventional tissue expansion (control) or with application Blossom Smart Expander Technology (intervention) in the first stage reconstruction (tissue expansion).

The intervention group involves the placement of the Mentor Spectrum tissue expander coupled with Blossom Syringe Assist device. The postoperative follow-up and subsequent surgery to exchange the device to a permanent implant is normal part of standard care.

A Mentor Spectrum adjustable saline breast implant for expansion, coupled with the Blossom Syringe Assist device, will be inserted above the pectoralis major muscle in the usual fashion. The nature of the surgery remains identical to that employed for conventional breast tissue expander insertion for reconstruction or augmentation.

Postoperative follow-up will occur within 1 week of surgery. Weekly follow-ups with documentation of clinical data throughout will also take place until completion of the expansion, stabilization of surgical scars, and removal of all percutaneous drains. Thereafter, follow-ups will be scheduled as needed (monthly) according to usual clinical practice in implant-based breast reconstruction in preparation for the second stage expander to definitive implant exchange.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 18 or older; pursuing non-oncologic breast reconstruction or augmentation; and ability to understand and the willingness to sign a written informed consent document (english language). Only patients desiring 2-staged tissue expander/ implant-based breast reconstruction will be approached for potential enrollment in the study.

Exclusion Criteria:

* Patients with active breast cancer; recent steroid use; major medical comorbidities (defined as ASA III or greater); a connective tissue disorder; are pregnant or nursing; are unable to understand and sign the english language consent forms; or age over 65 years, will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Time until completion of tissue expansion | Expansion is expected to be completed between 3 and 6 months after the stage 1 surgery.
  The time between placement of the tissue expander (stage 1 surgery) and completion of tissue expansion will be recorded and compared between each study arm.
Incidence of complications | Monitoring for complications will occur until removal of the tissue expander device during the second stage surgery (approximately 6 months)
  Any occurrence of surgical complications, such as infection, seroma, hematoma, extrusion, wound breakdown, and/ or device malfunction, etc. will be monitored and recorded in each study arm.

SECONDARY OUTCOMES:
Patient satisfaction (BreastQ) | Survey responses will be collected at standard post-operative time points (e.g. during each post-operative visit; 1 week, 3 weeks, 6 weeks post-op) until the second stage surgery (3 to 6 months).
  Patient satisfaction will be assessed using the validated BreastQ survey.
Patient satisfaction (device specific survey) | Survey responses will be collected at standard post-operative time points (e.g. during each post-operative visit; 1 week, 3 weeks, 6 weeks post-op) until the second stage surgery (3 to 6 months).
  Patient satisfaction will be assessed using a device-specific survey.
Pain associated with tissue expansion | Patient pain will be assessed routinely (e.g. during each post-operative visit; 1 week, 3 weeks, 6 weeks post-op) until tissue expansion is complete (3 to 6 months).
  Pain will be assessed using a study-specific survey.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Hospital and Clinics, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No